CLINICAL TRIAL: NCT02974803
Title: A Phase II Study of Concurrent Dabrafenib and Trametinib With Stereotactic Radiation in the Management of Patients With BRAF Mutation-Positive Malignant Melanoma and Brain Metastases
Brief Title: Concurrent Dabrafenib + Trametinib With Sterotactic Radiation in BRAF Mutation-Positive Malignant Melanoma and Brain Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Very slow accrual
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I224
Record Dates: First submitted 2016-11-23; First posted 2016-11-28 (Estimated); Results first posted 2021-08-17 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-07

CONDITIONS: Melanoma; Brain Metastases
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dabrafenib and Trametinib (Experimental): Dabrafenib, PO, 150mg BID Continuously Trameteinib, PO 2mg OD Continuously
  Interventions: Drug: Dabrafenib; Drug: Trametinib

INTERVENTIONS:
Drug: Dabrafenib — Dabrafenib 150 mg twice a day until progression or unaccepted toxicity.
Drug: Trametinib — Trametinib 2 mg once daily until progression or unaccepted toxicity.

SUMMARY:
Dabrafenib and trametinib are drugs that are usually given for the treatment of melanoma. Combinations of dabrafenib and trametinib have also been studied and when used together have shown to increase tumour shrinkage in animals compared to either drug alone. Dabrafenib and trametinib have also shown potential to penetrate the blood-brain-barrier when given together and have an effect on brain metastases. Giving these drugs at the same time and then giving brain stereotactic radiosurgery (SRS) may also be preferred in patients with brain metastases

DETAILED DESCRIPTION:
The purpose of this study is to find out the effects of giving dabrafenib in combination with trametinib continuously with stereotactic radiotherapy (SRS) has on melanoma and brain metastases.

Stereotactic Radiosurgery (SRS) is a non-surgical radiation therapy used to treat tumours of the brain. It can deliver precisely targeted radiation. Currently SRS alone is the usual treatment for patients with up to 4 brain lesions. This study will include 2 groups 1) patients with 1-4 brain lesions treated with SRS concurrently with dabrafenib and trametinib and 2) patients with 5-10 brain lesions treated with SRS concurrently with dabrafenib and trametinib.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed melanoma metastatic to brain and determined to be BRAF V600 mutated.
* Age ≥ 18 years.
* Karnofsky Performance Status of 70-100 (Appendix I).
* Patients must have a life expectancy of at least 12 weeks.
* Presence of measurable disease (i.e. present with at least one measurable CNS lesion per RECIST 1.1).
* Presence of 1-10 brain metastases as confirmed on a thin slice axial T1 post-gadolinium MRI sequence. The maximum diameter of a single brain lesion should be ≤ 4 cm and presence of a measurable lesion ≥ 1cm based on baseline MRI of brain.
* All CNS metastases amenable to single fraction SRS and or fractionated SRS. Hemorrhagic lesions are allowed if the treating radiation oncologist deems the lesion amenable to focal SRS.
* Able to swallow and retain oral medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* Laboratory requirements (within 14 days prior to registration):

  * ANC ≥ 1.2 x 10^9/L
  * Hemoglobin ≥ 90 g/L
  * Platelet count ≥ 100 x 10^9/L
  * PT/INR & PTT ≤ 1.3 x ULN
  * Total bilirubin ≤ 1.5 x ULN
  * AST and ALT ≤ 2.5 x ULN
  * Serum creatinine or ≤ 1.5 x ULN or Creatinine Clearance ≥ 50 ml/min (calculated by Cockcroft and Gault)
  * LVEF ≥ LLN (within 28 days prior to registration)
  * No prior treatment with a BRAF inhibitor or MEK inhibitor.
  * No known ocular or primary mucosal melanoma.
  * No prior systemic anti-cancer treatment within the last 2 weeks preceding the frist dose of dabrafenib and trametinib. Patients must have recoved from clinical manifestations of toxicity related to prior systemic therapy and have adequate washout as follows: Longest of one of the following:

    * two weeks
    * 5 half-lives for investigational agents
    * Standard cycle length of standard therapies
  * Prior systemic treatment in the adjuvant setting is allowed.
  * No current use of a prohibited medication as described in section 7.2.
  * No history of malignancy with confirmed activating RAS mutation at any time.
  * No history of malignancy other than disease under study within 3 years of study enrollment.
  * No leptomeningeal metastases or metastases causing spinal cord compression that are symptomatic or untreated or not stable for ≥ 3 months. Subjects on stable dose of corticosteroids > 2 weeks or who have been off of corticosteroids for at least 2 weeks can be enrolled with approval of CCTG.
  * No serious or unstable pre-existing medical conditions, psychiatric disorders or other conditions that could interfere with the subject's safety, obtaining informed consent or compliance with study procedures.
  * No history of Hepatitis B Virus or Hepatitis C Virus infection
  * No history or evidence of cardiovascular risk No history or current eveidence/risk of retinal vein occlusion or central serous retinopathy
  * No known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study treatments, their excipients, and/or dimethyl sulfoxide.
  * No pregnant or lactating women.
  * No hisotry of interstitial lung disease or active pneumonitis.
  * Presence of any one brain metastases >4cm in maximal diameter, and/or presence of brain metastase of less than 1cm.
  * No prior whole brain radiation
  * No brainstem metastses
  * No contrindications to MRI and/or Gadolinimum contrast or sterotactic brain radiation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arjun Sahgal, Study Chair — Odette Cancer Centre, Toronto, ON Canada; Teresa Petrella, Study Chair — Odette Cancer Centre, Toronto, ON Canada
Locations (6):
- Canada (6):
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dabrafenib and Trametinib: Dabrafenib, PO, 150mg BID Continuously Trameteinib, PO 2mg OD Continuously
  Dabrafenib
  Trametinib
Period: Overall Study
Arm/Group | Dabrafenib and Trametinib
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dabrafenib and Trametinib
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 63 [27 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 6

OUTCOME MEASURES:

1. Primary Outcome: Intracranial Objective Response Rate
Time Frame: 24 months
Population: The study was closed early because of very slow accrual and no final analysis was performed because the collected data cannot be considered reliable since they were not verified, reviewed or cleaned.
Arm/Group | Dabrafenib and Trametinib
Number analyzed (Participants) | 0

2. Secondary Outcome: Extra-cranial Objective Response Rate
Description: Response will be assessed using RECIST v1.1
Time Frame: 24 months
Population: as for outcome 1
Arm/Group | Dabrafenib and Trametinib
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of Response
Description: Response will be assessed using RECIST v1.1
Time Frame: 24 months
Population: as for outcome 1
Arm/Group | Dabrafenib and Trametinib
Number analyzed (Participants) | 0

4. Secondary Outcome: Intracranial Progression Free Survival
Description: Response will be assessed using RECIST v1.1
Time Frame: 24 months
Population: as for outcome 1
Arm/Group | Dabrafenib and Trametinib
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Progression Free Survival
Description: Response will be assessed using RECIST v1.1
Time Frame: 24 months
Population: as for outcome 1
Arm/Group | Dabrafenib and Trametinib
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Overall Objective Response Rate
Description: Response will be assessed using RECIST v1.1
Time Frame: 24 months
Population: as for outcome 1
Arm/Group | Dabrafenib and Trametinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 24 months
Description: The study was closed early because of very slow accrual and no final analysis was performed because the collected data cannot be considered reliable since they were not verified, reviewed or cleaned.
Arm/Group | Dabrafenib and Trametinib
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-26): https://cdn.clinicaltrials.gov/large-docs/03/NCT02974803/Prot_SAP_000.pdf